CLINICAL TRIAL: NCT07136311
Title: Otoacoustics Emissions Contralateral Supression Test
Brief Title: The Effect of Obesity on Contralateral Suppression in Patients With Multiple Sclerosis
Acronym: MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Asuman Kucukoner, Principal Investigator, Ondokuz Mayıs University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Ethics number 2022/ 300
Record Dates: First submitted 2025-07-30; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis; Obesity; Hearing Loss
MeSH Terms: conditions — Multiple Sclerosis; Obesity; Hearing Loss

STUDY DESIGN:
Intervention Model Description: Interventional (Clinical Trial)
Masking Description: This is an observational study with no intervention; therefore, no masking was applied. All participants and investigators were aware of the group assignments (obese vs. non-obese), and no parties beyond those listed were masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obese and Non-Obese MS Patients Undergoing DPOAE Suppression Test (Other): Diagnostic Test, "DPOAE with Contralateral Suppression"
  Interventions: Diagnostic Test: DPOAE with Contralateral Suppression
- Non-Obese MS Patients (Other): Diagnostic Test - DPOAE with Contralateral Suppression
  Interventions: Diagnostic Test: DPOAE with Contralateral Suppression

INTERVENTIONS:
Diagnostic Test: DPOAE with Contralateral Suppression — Participants will undergo distortion evoked otoacoustic emissions (DPOAE) testing with contralateral broadband noise stimulation. The test is performed to evaluate auditory efferent system function, specifically the presence and degree of contralateral suppression. No medication or treatment is administered as part of the study. The procedure is non-invasive and commonly used in auditory diagnostics.

SUMMARY:
This study investigates how obesity may affect the auditory system in individuals with Multiple Sclerosis (MS). Specifically, it examines the brain's ability to process and suppress sounds (contralateral suppression).

The test is painless and brief. It provides information about the condition of the auditory nerve pathways. The goal is to better understand how obesity may influence this system and to improve follow-up and support for individuals with MS.

DETAILED DESCRIPTION:
This study investigates the potential impact of obesity on auditory efferent system function in individuals diagnosed with Multiple Sclerosis (MS). Specifically, it focuses on assessing contralateral suppression of Distortion Product Otoacoustic Emissions (DPOAEs), a non-invasive, objective method for evaluating the integrity of the cochlear outer hair cells and the medial olivocochlear (MOC) efferent system.

Participants will undergo a brief and painless auditory test, during which DPOAEs are recorded both in quiet and with contralateral acoustic stimulation. This approach allows for the assessment of the brainstem's ability to suppress cochlear responses, which reflects central auditory processing capabilities.

By comparing suppression patterns across participants with different body mass index (BMI) classifications, the study aims to identify whether obesity contributes to functional changes in the auditory efferent system among MS patients.

The outcomes of this research may enhance the understanding of how metabolic factors such as obesity interact with neurological conditions like MS, potentially guiding more personalized clinical monitoring and interventions.

ELIGIBILITY:
Eligibility Criteria Minimum Age: 18 Years Maximum Age: 50 Years Sex: All Gender Based: No Accepts Healthy Volunteers: No

Inclusion Criteria:

Ability to cooperate with the applied scales and auditory tests

Normal findings in otoscopic examination (ear, nose, and throat evaluation)

Absence of any neurological, psychiatric, or metabolic disease other than Multiple Sclerosis (MS)

No history of significant noise exposure

For female participants: not pregnant and not in the menstrual period

Exclusion Criteria:

Presence of active middle ear pathology (e.g., otitis media, tympanic membrane perforation)

Abnormal tympanometric findings

Hearing loss exceeding 20 dB HL at any frequency between 500-4000 Hz

Neurological or psychiatric disorders other than MS

History of ear surgery or otologic trauma

Use of medications known to affect auditory function (e.g., ototoxic drugs)

Inability to cooperate with audiological testing

Pregnancy

Diagnosis of metabolic or endocrine disorders (e.g., uncontrolled diabetes, thyroid dysfunction)

Body Mass Index (BMI) below 18.5 (underweight) or above 40 (morbid obesity)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Contralateral supression | Within 12 months of MS diagnosis
  Comparison of contralateral suppression values of distortion product otoacoustic emissions (DPOAEs) between obese and non-obese patients with Multiple Sclerosis (MS) at multiple frequencies (1 kHz, 1.4 kHz, 2 kHz, 2.8 kHz, 4 kHz, 5.6 kHz, and 8 kHz).

SECONDARY OUTCOMES:
DPOAE Amplitude Levels | Within 12 months of MS diagnosis
  Evaluation and comparison of baseline DPOAE amplitudes (without contralateral stimulation) between obese and non-obese MS patients at all test frequencies (1 kHz, 1.4 kHz, 2 kHz, 2.8 kHz, 4 kHz, 5.6 kHz, and 8 kHz).

CONTACTS AND LOCATIONS:
Overall Officials: Asuman Küçüköner, PD Dr, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data sharing is not planned prior to the publication of the study. Access may be considered after publication, upon request and subject to ethical approval.

REFERENCES:
- [Background] Kucukoner A, Kucukoner O, Ozgur A, Terzi M. Effect of Medial Olivocochlear Efferents on Speech Discrimination in Noise in Multiple Sclerosis. Noise Health. 2024 Oct-Dec 01;26(123):507-513. doi: 10.4103/nah.nah_71_23. Epub 2024 Dec 30. PMID 39787552

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT07136311/Prot_SAP_000.pdf